CLINICAL TRIAL: NCT05831384
Title: Does Diabetes Related Distress Impact on Balance Glycemic ?
Acronym: DDS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230419; 2023-A00342-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Diabetes
Keywords: Diabetes; Distress
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to assess the overall diabetes distress score in adult patients with diabetes during their hospitalization in a diabetes ward, using the Diabetes Distress Scale (DDS-17).

The correlation between the overall diabetes distress score and the patient's glycosylated haemoglobin will then be assessed.

DETAILED DESCRIPTION:
The health consequences of emotional problems are associated with poor self-care behaviour, poor metabolic outcomes (HbA1c) and reduced quality of life. If quarterly glycated haemoglobin (HbA1c) testing is the gold standard for monitoring the risk of diabetes complications, should it not be systematically combined with the assessment of distress related to living with diabetes? To our knowledge, there are few studies in France that have correlated glycaemic control with a scale assessing the emotional stress factors associated with diabetes.

The main objective is to evaluate diabetes-related distress in adult patients with diabetes during their hospitalization in a diabetes ward, using a self-assessment instrument: the Diabetes Distress Scale (DDS-17).

The secondary objective is to assess the correlation between the overall diabetes distress score and the patient's glycosylated haemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Patients living with type 1 or type 2 diabetes.
* Patients hospitalised in the diabetes department of the IE3M.
* Patients aged ⩾ 18 years.
* Patients agreeing to participate in this study after information.
* Beneficiary of the health insurance.

Exclusion Criteria:

* Refusal to participate.
* Inability to communicate in French.
* Inability to read or write French.
* Communication disorders.
* History of psychiatric disorders, dementia.
* Patient under guardianship or curatorship.
* Patient not affiliated to social security.
* Patient affiliated to the Aide Médicale d'Etat (AME).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult hospitalized patients for diabetes at IE3M.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Overall diabetes distress score | at baseline
  The primary endpoint is the overall diabetes distress score obtained by the DDS-17 psychometric tool. Each item is rated on a 6-point scale ranging from (1) "not a problem" to (6) "a very significant problem".
  Each of the 17 criteria of the DDS17 is rated on a 6-point scale ranging from (1) "not a problem" to (6) "a very important problem".
  The scale gives an overall distress score based on the average responses on the 1-6 scale for the 17 items.
  Interpretation of the DDS 17 total scores:
  * Mean score < 2.0 = reflects little or no distress
  * Mean score between 2.0 and 2.9 = reflects moderate distress
  * Mean score > 3.0 = reflects high distress.

SECONDARY OUTCOMES:
The The patient's glycated haemoglobin (Hba1c) result, expressed as a %, taken during the standard check-up on the day of admission to hospital result (Hba1c) | at baseline
  The patient's glycated haemoglobin (Hba1c) result, expressed as a %, taken during the standard check-up on the day of admission to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Alvitre, Nursing degree, Principal Investigator — Diabetology department - Hospital of Pitié Salpêtrière
Locations (1):
- Diabetology department - Hospital of Pitié Salpêtrière - APHP, Paris, France